CLINICAL TRIAL: NCT04523246
Title: Training the Innate Immune System Against SARS-COV-2 (COVID-19) Using the Shingrix Vaccine in Nursing Home Residents: A Randomized, Doubled-Blinded, Comparative Group Observational Study
Brief Title: Training the Innate Immune System Against SARS-CoV-2 (COVID-19) Using the Shingrix Vaccine in Nursing Home Residents
Acronym: NH-Shingrix
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma Medical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 12394
Record Dates: First submitted 2020-08-20; First posted 2020-08-21 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Herpes Zoster; Allergy and Immunology; Corona Virus Infection
Keywords: Herpes Zoster; corona virus infection; allergy and immunology
MeSH Terms: conditions — Herpes Zoster; Hypersensitivity; Coronavirus Infections | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Two hundred nursing home residents, both men and women, aged >65 years, who have not acquired COVID-19 (verified through a screening questionnaire and by both viral antigen and antibody testing at the screen and least one week before the first injection) will get two intramuscular injections containing either the Shingrix vaccine, and the other half, two injections containing a normal saline (comparison) approximately two months apart. Blood samples are collected before the baseline injection (day zero), 1 day after the second injection (61 days post) and 1 month following the second injection (90 days). Weekly symptom checks and monthly antibody testing around day 180- will identify residents with COVID-19 and the severity of COVID-19 symptoms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding is done to ensure staff and residents do not modify reports or reporting of COVID symptoms and to minimize other behaviors (such as sleeping, eating habits, physical activity) that may affect their innate immune system. It will also serve to minimize any bias in the processing/analysis of samples and the interpretation of the study results.
  During the conduct of the study, only three people (the statistician and 2 research nurses who will reconstitute, draw up, and administer the injections) will have knowledge of the group assignments. Participants, the staff at the nursing home, the staff collecting the COVID symptom data, and study investigators are blinded to the subject assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Shingrix (Experimental): Shingrix Dosage: two .5 ml injections into the deltoid muscle, administered 3 months apart (Day 0 and Day 90).
  Interventions: Biological: SHINGRIX (Zoster Vaccine REcombinant, Adjuvanted)
- Normal Saline (Placebo Comparator): Sterile Normal Saline Solution, two .5 ml injections into the deltoid muscle, administered 3 months apart (Day 0 and Day 90)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Biological: SHINGRIX (Zoster Vaccine REcombinant, Adjuvanted) — The Shingrix vaccine is a subunit vaccine that contains the recombinant varicella zoster virus (VZV) glycoprotein E (gE), adjuvanted with the proprietary Adjuvant System (AS01B). The AS01B Adjuvant system consists of two immune-stimulants, the saponin, Quillaja saponaria Molina, fraction 21 (QS21), and the toll-like receptor 4 (TLR4) agonist, MPL (3-O-desacyl-40-MPL) that enhance the release of interferon gamma (IFNϒ), which in turn stimulates activation and recruitment of blood monocyte-derived and resident lymph node dendritic cells to take up and present gE to cluster of differentiation 4 (CD4+) T cells.
  Other Names: Zoster Vaccine Recombinant, Adjuvanted
  Arms: Shingrix
Drug: Normal Saline — Sterile normal saline, inactive control.
  Other Names: saline
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to measure the effect of the Shingrix vaccine on your immune system and whether that has any effect on the body's ability to fight off other infections such as COVID-19. We hypothesize that:

H1: Shingrix vaccination will elevate acute and trained immunity

H2: For 6 months following the first injection, increased levels of acute and trained immunity is associated with less disease, including fewer hospitalizations and deaths associated with flu, pneumonia, and COVID-19.

DETAILED DESCRIPTION:
The purpose of this pilot study is to provide preliminary data in support of the concept that training of the innate immune system occurs following immunization (2 doses ,3 months apart) with the Shingrix vaccine as compared to placebo (normal saline) in older adults residing in nursing homes. Two hundred nursing home residents, both men and women, aged >65 years, who have not acquired COVID-19 (verified through a screening questionnaire and by both viral antigen and antibody testing at the screen and least one week before the first injection) will get two intramuscular injections containing either the Shingrix vaccine, and the other half, two injections containing a normal saline (placebo comparison) approximately three months apart. Blood samples are collected before the baseline injection (day zero), 1 day after the second injection (91 days post) and 1 month following the second injection (120 days). Weekly symptom checks and monthly antibody testing around day 180- will identify residents with COVID-19 and the severity of COVID-19 symptoms.

The primary outcome is the difference in immune cell capacity to produce type I interferon, interferon associated molecules, and proinflammatory mediators after receiving a 2 injection series of the Shingrix vaccine versus normal saline. Secondary outcomes include differences in hospitalization, pulmonary infections, and positive COVID-19 cases (via antibody testing on days 90, 120, and 180) in the Shingrix and normal saline groups. We anticipate that residents receiving the Shingrix vaccine will demonstrate signs of "trained" immunity compared to a control group receiving saline injections.

ELIGIBILITY:
Inclusion Criteria:

1. Meet Centers for Medicare and Medicaid definition for Long term care resident.
2. 65 years and older.
3. Have already received or provide consent to receive the 2020 flu vaccine.
4. Negative screen (within the last 2 weeks) for COVID 19 virus.
5. Has a history of chickenpox or shingles.
6. Able to read and speak English.
7. Able to provide informed consent and assent (with guardian/health care proxy).

Exclusion Criteria:

1. Brief Interview of Mental Status (BIMS) score <8 (indicating severe dementia).
2. Prior vaccination with the Shingrix.
3. Positive test for COVID 19 or prior history of COVID 19 infection.
4. Conditions that confound the interpretation of the innate immune measures. (i.e. Terminal condition, receiving hospice, Stage 3 and 4 open wound, Chemotherapy, immune modulators or other immunosuppressants, autoimmune disorders, and BMI < 20 kg/m2).
5. Conditions that confound interpretation of respiratory symptoms. (i.e Ventilator dependent, receiving more that 2-3 liters/min of oxygen by nasal cannula, chronic diarrhea, recurrent infections).

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 217 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Evidenced of active and trained innate immunity | Day 91 and 120 (post vaccination)
  The primary outcome is change in the release of Type I interferon, interferon gamma, interferon associated molecules, and proinflammatory mediators released from monocytes/macrophages and natural killer cells (including gene activation) after receiving 2 injections of the Shingrix vaccine versus normal saline.

SECONDARY OUTCOMES:
Respiratory Disease Severity (6 month) | Days 120 through 180
  cases ( nasal swab for viral antigen and antibody testing), symptoms (symptom checklist), hospitalizations (MDS 3.0 report/chart reviews) and deaths (MDS 3.0 report/chart reviews) associated with flu, pneumonia, and COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara W. Carlson, RN, Ph.D., Study Director — Professor, University of Oklahoma Health Sciences Center
Locations (1):
- Fran and Earl Ziegler College of Nursing, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No